CLINICAL TRIAL: NCT05331703
Title: Virtual Reality Versus Mirror Therapy on Balance and Muscle Strength in Children With Hemiplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, samar salem, assistant professor at faculty of physical therapy at October 6 university, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/0035A342
Record Dates: First submitted 2022-03-28; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): will receive a designed physical therapy program in addition to program of virtual reality
  Interventions: Other: designed physical therapy program in addition to program of virtual reality.
- group B (Experimental): will receive a designed physical therapy program in addition to program of mirror therapy.
  Interventions: Other: designed physical therapy program in addition to program of mirror therapy.

INTERVENTIONS:
Other: designed physical therapy program in addition to program of virtual reality. — physical therapy program in addition to program of virtual reality.
  Arms: group A
Other: designed physical therapy program in addition to program of mirror therapy. — physical therapy program in addition to program of mirror therapy.
  Arms: group B

SUMMARY:
Previous research has demonstrated balance deficits ranging from 28%-43% depending on the nature of the balance task in individuals with CP compared to controls (Kenis-Coskun et al., 2016). As balance is critical for underlying normal movement, improvements in static and dynamic balance are important goals in rehabilitation for ambulatory children with CP (Saether et al., 2013).

Balance deficits are among the symptoms that having a more profound impact on motor function and quality of life inn with CP children (Lai et al., 2017). Poor balance reduces the ability to perform gait-related activities and increases the risk of falling, which, in turn, limits participation in daily activities, including sports and physical activities (Usuba et al., 2015).

ELIGIBILITY:
Inclusion Criteria:

* Their ages will range from 6 to 10 years old.
* The degree of spasticity will range from 1+ to 2 grades according to Modified Ashworth scale (NUMANO and Günel, 2011) (Appendix II).
* They will be on level I and II on Gross Motor Function Classification System (GMFCS) (Palisano et al., 2008) (Appendix III).
* Their heights will be one meter or more.
* They will be able to follow the verbal commands or instructions.

Exclusion Criteria:

* Severe visual or auditory problems.
* Epilepsy.
* History of surgical interference in lower limbs.
* Botulinum toxin injections of the lower limbs during the previous six

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-12-22 (Estimated); Primary Completion 2023-03-22 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Biodex balance system | 3 months
  The Biodex balance System to measures postural stability under dynamic stress.
Hand held dynamometer | 3 months
  The hand held dynamometry to measure muscle strength of non-disabled children

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Eldin, Cairo, October, Egypt